CLINICAL TRIAL: NCT00421161
Title: Phase 1 and 2 Study on the Efficacy and Side Effects of Olive Oil and Omega 3 Local Treatment in Stasis Dermatitis
Brief Title: Olive Oil With Omega 3 to Treat Stasis Dermatitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Refael Segal
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Dermatitis
Keywords: olive oil; stasis dermatitis; Patients with stasis dermatitis for at least six months.
MeSH Terms: conditions — Dermatitis | interventions — Olive Oil; Docosahexaenoic Acids

INTERVENTIONS:
Drug: olive oil and omega 3 in a combined cream

SUMMARY:
Olive oil and Omega 3 have many anti inflammatory effects that may be beneficial in the inflammation and edema of chronic stasis dermatitis. The olive oil contains many mono unsaturated fatty acids and anti oxidants that may add to the well being of a diseased skin by improving cell membrane homeostasis.

DETAILED DESCRIPTION:
Patients with chronic stasis dermatitis due to venous insufficiency will be treated with the study cream and as control we will use "Venoroutone" . Patients will be followed weekly at the clinic of the vascular surgery at Assaf Harofeh MC.

ELIGIBILITY:
Inclusion Criteria:

* Patints with stasis dermatitis for 6 months at least

Exclusion Criteria:

* skin ulceration or infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2007-01; Study Completion 2007-03

PRIMARY OUTCOMES:
improvement in subjective and objective skin changes of patient: pain, edema, redness, size of involement,

CONTACTS AND LOCATIONS:
Overall Officials: Arie Bass, MD, Principal Investigator — Assaf Harofe MC
Locations (3):
- Israel (3):
  - Assaf Harofe MC, Ẕerifin, Beer Yaacov
  - Clinic of vascular surgery, Assaf Harofe MC, Ẕerifin, Zerifin
  - Clinic of Vascular Surgery, Ẕerifin, Zerifin

REFERENCES:
- [Background] Sapino S, Carlotti ME, Peira E, Gallarate M. Hemp-seed and olive oils: their stability against oxidation and use in O/W emulsions. J Cosmet Sci. 2005 Jul-Aug;56(4):227-51. PMID 16130045